CLINICAL TRIAL: NCT03078140
Title: The Study to Compare Iodine Supplement Strategies Between Routine Iodine Supplementation and Selective Iodine Supplementation
Brief Title: Iodine Supplement Strategies Between Routine Iodine Supplementation and Selective Iodine Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kuntharee Traisrisilp, Principle Investigator, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4298
Record Dates: First submitted 2017-02-27; First posted 2017-03-13 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Pregnancy Related; Iodine Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triferdine (Active Comparator): Triferdine 1 tablet by mouth daily. Start after 1st trimester until delivery
  Interventions: Dietary Supplement: Triferdine
- Triferdine/Ferli-6 (Active Comparator): Triferdine or ferli-6 1 tablet by mouth daily base on iodine status. The supplement will give after 1st trimester until delivery
  Interventions: Dietary Supplement: Triferdine/Ferli-6

INTERVENTIONS:
Dietary Supplement: Triferdine — Triferdine 1 tablet daily Start from 14 weeks of gestation until delivery
  Arms: Triferdine
Dietary Supplement: Triferdine/Ferli-6 — For the participants assigned to this group, urine iodine level will be checked first.
  For participants with normal urine iodine level, Ferli-6 1 tab daily will be given.
  For those with low urine iodine level, Triferdine 1 tab daily will be given. Medication will be started from 14 weeks of gestation until delivery.
  Arms: Triferdine/Ferli-6

SUMMARY:
Pregnant women who attend at our antenatal clinic will random to 2 groups. First will receive routine iodine supplementation. The other will receive iodinated pill or only iron supplementation base on their urine iodine status.

ELIGIBILITY:
Inclusion Criteria:

* first visit for antenatal care in the first trimester
* singleton pregnancy
* delivered at Maharaj Nakorn Chiangmai Hospital

Exclusion Criteria:

* thyroid disease which diagnosed before pregnancy or currently
* history of thyroid gland surgery or iodine ablation therapy
* received iodine supplement before pregnancy
* received any medication for thyroid disease treatment, within 6 weeks postpartum women or breast feeding period
* family history of thyroid disease
* having underlying disease or contraindication which cannot received iodine supplement
* loss follow-up or incomplete data.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
iodine status | at delivery
  mean urine iodine

CONTACTS AND LOCATIONS:
Locations (1):
- Kuntharee Traisrisilp, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No